CLINICAL TRIAL: NCT00603252
Title: Evaluate the Effect of Risk Factors That Influence the Immunogenicity of GSK Biologicals' Twinrix Compared to Hepatitis A and Hepatitis B Vaccines Given Separately and to Show the Non-inferiority Between the Vaccines in Adults
Brief Title: Study to Show That the Combined Hepatitis A and B Vaccine is Non-inferior to Monovalent Vaccines in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111149
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis B; Hepatitis A
Keywords: combined hepatitis A and B vaccine; risk factors
MeSH Terms: conditions — Hepatitis B; Hepatitis A | interventions — twinrix; Engerix-B; Hepatitis A Vaccines; Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Twinrix
Biological: Engerix-B
Biological: Havrix
Biological: HBVAXPRO
Biological: Vaqta

SUMMARY:
This protocol posting describes the booster phase of the study. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT number = NCT00289731).

DETAILED DESCRIPTION:
All subjects will receive a dose of the vaccine that they received in the primary study (100382), approximately 4 years after the first dose. Blood samples will be taken before and after the administration of the vaccine dose to evaluate the anti-HAV and anti-HBs antibody response.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* A male or female who completed the primary vaccination phase of the study.
* Written informed consent obtained from the subject.
* If the subject is female, she must be of non-childbearing potential, or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* History of any hepatitis A or hepatitis B vaccination or infection, since the primary vaccination study.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrolment.
* Pregnant or lactating female.

Min Age: 41 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Anti-HAV immune response to the challenge dose
Anti-HBs antibody response to the challenge dose

SECONDARY OUTCOMES:
Percentage of subjects with anti-HAV antibody titres ≥ 15 mIU/ml and GMTs calculated on seropositive subjects | Two weeks and one month after the challenge dose
Percentage of subjects with anti-HBs antibody titres ≥ 3.3 mIU/ml, ≥ 10 mIU/ml, ≥ 100 mIU/ml and anti-HBs GMTs calculated on seropositive subjects | Two weeks and one month after the challenge dose
Occurrence and intensity of solicited local symptoms | In the 4-day follow-up period after the challenge dose
Occurrence, intensity and relationship of solicited general symptoms | In the 4-day follow-up period after the challenge dose
Occurrence, intensity and relationship to vaccination of unsolicited symptoms reported | During the 31-day follow-up period after the challenge dose
Occurrence of all serious adverse events (SAEs) reported | Following the administration of the challenge dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- GSK Investigational Site, Wilrijk, Belgium
- Germany (7):
  - GSK Investigational Site, Finsterwalde, Brandenburg
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Geringswalde, Saxony
  - GSK Investigational Site, Pirna, Saxony
  - GSK Investigational Site, Bad Bramstedt, Schleswig-Holstein
  - GSK Investigational Site, Bad Segeberg, Schleswig-Holstein
  - GSK Investigational Site, Elmshorn, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Chlibek R, von Sonnenburg F, Van Damme P, Smetana J, Tichy P, Gunapalaiah B, Leyssen M, Jacquet JM. Antibody persistence and immune memory 4 years post-vaccination with combined hepatitis A and B vaccine in adults aged over 40 years. J Travel Med. 2011 Mar-Apr;18(2):145-8. doi: 10.1111/j.1708-8305.2010.00499.x. Epub 2011 Feb 7. PMID 21366801
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 111149 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111149 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111149 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111149 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111149 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register